CLINICAL TRIAL: NCT05726136
Title: Comparison of Albumin and Ringer's Solution for Optimization of the Plasma Volume and Hemodynamics During Laparoscopic Surgery.
Brief Title: Fluid Challenge and Plasma Volume, During Surgery
Acronym: FC-VE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Joachim Zdolsek (Other)
Responsible Party: Sponsor-Investigator, Joachim Zdolsek, consultant, assoc prof, University Hospital, Linkoeping
Organization: University Hospital, Linkoeping (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FC-VE
Record Dates: First submitted 2023-01-15; First posted 2023-02-13 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Colorectal Cancer; Urologic Cancer; Gynecologic Cancer; Colorectal Disorders; Benign Neoplasm
Keywords: laparoscopic surgery, fluid therapy, plasma volume
MeSH Terms: conditions — Colorectal Neoplasms; Urologic Neoplasms; Neoplasms | interventions — Ringer's acetate; zidovudine 5'-monophosphate-mannose-albumin conjugate; Albumins; galactosamine-conjugated serum albumin-conjugated-(rhodamine X)20

STUDY DESIGN:
Intervention Model Description: 3 randomized parallel groups, with 20 patients in each group. Each group receives a prespecified fluid regime with: 1. acetated Ringers 2. albumin 5% or 3. albumin 20%
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- acetated Ringers (Experimental): The circulatory effect of a bolus infusion with 4 ml/kg body weight of acetated Ringers will be studied. If cardiac output increase with 10% a second bolus will be infused and further studied.
  Interventions: Drug: acetated Ringers
- albumin 5% (Experimental): The circulatory effect of a bolus infusion with 4 ml/kg body weight of Albumin 5% will be studied. If cardiac output increases with 10% a second bolus will be infused and further studied.
  Interventions: Drug: albumin 5%
- albumin 20% (Experimental): The circulatory effect of a bolus infusion with 1 ml/kg body weight of Albumin 20% will be studied. If cardiac output increase with 10% a second bolus will be infused and further studied.
  Interventions: Drug: albumin 20%

INTERVENTIONS:
Drug: acetated Ringers — After insufflation of carbon dioxide during an abdominal laparoscopic procedure, the first fluid bolus is infused. Circulatory and volume effects are studied. If cardiac output increase a second bolus is infused and studied.
  Other Names: Ringer's acetate; ringer acetate; acetate Ringer´s
  Arms: acetated Ringers
Drug: albumin 5% — After insufflation of carbon dioxide during an abdominal laparoscopic procedure, the first bolus of fluid is infused. Circulatory and volume effects are studied. If cardiac output increases a second bolus is infused and studied.
  Other Names: Albumin (Human) 5%; Human Albumin 5%
  Arms: albumin 5%
Drug: albumin 20% — After insufflation of carbon dioxide during an abdominal laparoscopic procedure, the first bolus of fluid is infused. Circulatory and volume effects are studied. If cardiac output increases a second bolus is infused and studied.
  Other Names: Human Albumin 20%; Albumin (Human) 20%
  Arms: albumin 20%

SUMMARY:
A short bolus infusion of fluid, called "fluid challenge" is commonly recommended for fluid treatment during longer surgery. However a prolonged increase of the blood volume is a prerequisite to recommend the technique. The purpose with the study is to examine the plasma expanding effect of three different fluid challenge strategies (acetated Ringers 4 ml/kg body weight, albumin 5% 4 ml/kg body weight or albumin 20% 1 ml/kg body weight), using hemoglobin as a dilution indicator.

DETAILED DESCRIPTION:
60 patients scheduled for laparoscopic abdominal surgery, with a duration exceeding 90 minutes will be included in the study. These are randomized to three different groups (20 in each groups): The first group of patients will receive boluses of acetated Ringers 4 ml/kg body weight. The second albumin 4 ml/kg body weight and the third group albumin 20% 1 ml/kg body weight.

Hemoglobin, albumin and colloid osmotic pressure (COP) is sampled the day before surgery and in the morning directly prior to the anesthesia. Bioimpedance, urine osmolality and urine-creatinin are also measured. After induction of surgery a Cardio Q probe is inserted threw the nose into the esophagus, for circulatory measurements. Initial/baseline blood samples are taken after insufflation of carbon dioxide to the abdomen. Before every bolus of fluid and 5, (10), 15, 20, 30, 40, (50) and (60) minutes new blood samples are taken for determination of hemoglobin, albumin and COP. Artery blood gases are sampled 15 minutes after every infusion or depending on the clinical need.

ELIGIBILITY:
Inclusion Criteria:

* Written consent to participate in the study
* For women: relevant contraceptive, menopausal or a negative pregnancy test.
* ASA category I to III
* Laparoscopic abdominal surgery, with a duration of at least 90 minutes.
* 18 to 80 years

Exclusion Criteria:

* Patients with known cardiac failure
* <18 or >80 years
* known allergy to albumin
* extracellular hyperhydration or hypervolemia
* kidney failure
* pregnancy or planned pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Plasma volume expansion after a fluid bolus | 60 minutes after an intravenous fluid bolus
  Plasma volume using hemoglobin as an indicator of dilution

SECONDARY OUTCOMES:
Fluid Balance | 18 to 24 hours
  Calculations of fluid balance
Stroke Volume | 60 minutes after an intravenous fluid bolus
  Change in stroke volume, measured with Cardio Q (oesophageal Doppler monitoring (ODM))
Arterial Blood Pressure | 60 minutes after an intravenous fluid bolus
  Mean Arterial Pressure, measured with an arterial line.
Heart Rate | 60 minutes after an intravenous fluid bolus
  Heart rate, measured with ECG and pulseoximeter.
Bioimpedance | 18 to 24 hours
  Bioimpedance measures, resistance and impedance converted to volume of body fluid compartments.
Serum Creatinin | 18 to 24 hours
  Serum Creatinin as a measure of kidney function
arterial pH | 60 minutes after an intravenous fluid bolus
  Influence of a fluid bolus on arterial blood gases
arterial Base Excess | 60 minutes after an intravenous fluid bolus
  Influence of a fluid bolus on arterial blood gases
arterial serum sodium | 60 minutes after an intravenous fluid bolus
  Influence of a fluid bolus on Sodium concentration
arterial serum chloride | 60 minutes after an intravenous fluid bolus
  Influence of a fluid bolus on Chloride concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Zdolsek, MD PhD, Principal Investigator — Department of Biomedical and Clinical Sciences, Linköping University, Linköping, Sweden
Locations (1):
- Vrinnevi Hospital, Norrköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: No
Individual de-identified results will be shared, when results are published.

DOCUMENTS (2):
  • Study Protocol (2022-07-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT05726136/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT05726136/SAP_001.pdf